CLINICAL TRIAL: NCT03040440
Title: Comparison of the Cuff Pressure of TaperGuard Endotracheal Tube and Cylindrical- Endotracheal Tube During Laparoscopic Surgery
Brief Title: Comparison of the Cuff Pressure of TaperGuard and Cylindrical- Endotracheal Tube During Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: KNUH 2016-03-001-004
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Cuff Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cylindrical endotracheal tube (Active Comparator): Cylindrical endotracheal tube was intubated in 32 participants
  Interventions: Device: Cylindrical endotracheal tube
- TaperGuard endotracheal tube (Experimental): TaperGuard endotracheal tube was intubated in 32 participants
  Interventions: Device: TaperGaurd endotracheal tube

INTERVENTIONS:
Device: Cylindrical endotracheal tube — Cylindrical endotracheal tube was intubated
  Arms: Cylindrical endotracheal tube
Device: TaperGaurd endotracheal tube — TaperGaurd endotracheal tube was intubated
  Arms: TaperGuard endotracheal tube

SUMMARY:
The purpose of this study was to compare the cuff pressure between cylindrical and TaperGuard endotracheal tube during laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Sixty four participants were assigned to one of the two groups: cylindrical and TaperGuard endotracheal tube. At the supine position, cuff pressure of endotracheal tube was measured before and after abdominal insufflation in the supine position. After insufflation the head-up position (30°) was made and cuff pressure was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were underwent laparoscopic cholecystectomy with American Society of Anesthesiologists physical status 1-3

Exclusion Criteria:

* history with respiratory disease, difficult intubation, and morbid obesity (body mass index more than 35 kg/m2).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
cuff pressure | 5 minutes after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, MD, Study Chair — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Yes